CLINICAL TRIAL: NCT03514342
Title: The Effects of Difference in Pupil Size Between Bilateral Eyes on Cardiac Sympathetic Nervous Activity Following Interscalene Brachial Plexus Block
Brief Title: The Effects of Horner's Syndrome Developing After Interscalene Brachial Plexus Block on Autonomic Nervous Activity
Status: Completed | Type: Observational
Sponsor: Daegu Catholic University Medical Center (Other)
Collaborators: Research Institute of Medical Science, Daegu Catholic University (Unknown)
Responsible Party: Principal Investigator, JongHae Kim, Associate Professor, Daegu Catholic University Medical Center
Other Study IDs: 2018-02
Record Dates: First submitted 2018-04-19; First posted 2018-05-02 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Brachial Plexus Block; Horner Syndrome; Autonomic Imbalance
Keywords: Heart rate variability; Mesopic pupil size
MeSH Terms: conditions — Horner Syndrome | interventions — Ropivacaine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Interscalene brachial plexus block: Ultrasound-guided interscalene brachial plexus block with 25 ml to 30 ml of 0.75% ropivacaine
  Interventions: Procedure: Interscalene brachial plexus block; Drug: 0.75% ropivacaine

INTERVENTIONS:
Procedure: Interscalene brachial plexus block — Under ultrasound guidance, the 5th to 7th cervical nerve roots are identified between anterior and middle scalene muscles and subsequently blocked.
Drug: 0.75% ropivacaine — Placement of 25 to 30 ml of 0.75% ropivacaine around the 5th to 7th cervical nerve roots
  Other Names: Naropin

SUMMARY:
This study evaluates the effects of Horner's syndrome on cardiac autonomic nervous activity after interscalene brachial plexus block. Cardiac autonomic nervous activity and bilateral pupil diameters will be measured in a scotopic light condition, 30 minutes after interscalene brachial plexus block under ultrasound guidance and 15 minutes after the subsequent sitting position.

DETAILED DESCRIPTION:
Stellate ganglia provide sympathetic fibers to the heart. Ipsilateral stellate ganglion block accompanied by interscalene brachial plexus block causes Horner's syndrome presenting with miosis, ptosis, and anhidrosis. The extent of Horner's syndrome can be represented by the difference in pupil diameter between bilateral eyes. Cardiac autonomic nervous activity affected by stellate ganglion block can be measured by calculation of heart rate variability parameters.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status 1
* Arthroscopic shoulder surgery under interscalene brachial plexus block

Exclusion Criteria:

* Coagulopathy
* Infection at the site of brachial plexus block
* Peripheral neuropathy or neurologic sequelae on the operative limb
* Allergy to local anesthetics or history of allergic shock
* Psychiatric diseases
* Patient refusal
* Difficulty communicating with medical personnel
* Arrhythmias
* Ischemic heart disease
* Hypertension
* Diabetes mellitus
* Thyroid dysfunction
* Conduction abnormalities on electrocardiogram
* Electrolyte imbalance
* Medications affecting cardiac conduction
* Contralateral vocal cord palsy
* Contralateral hemidiaphragmatic paresis or paralysis
* Contralateral pneumothorax or hemothorax

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Tertiary hospital
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Post-sitting sympathetic nervous activity | 15 minutes after the sitting position following interscalene brachial plexus block
  Natural-log transformed low frequency power of heart rate variability calculated using R wave to R wave intervals obtained for 5 minutes between 10 and 15 minutes after the sitting position following interscalene brachial plexus block

SECONDARY OUTCOMES:
Post-sitting ipsilateral pupil diameter | 15 minutes after the sitting position following interscalene brachial plexus block
  Ipsilateral pupil diameter measured under a mesopic condition 15 minutes after the sitting position following interscalene brachial plexus block
Post-sitting contralateral pupil diameter | 15 minutes after the sitting position following interscalene brachial plexus block
  Contralateral pupil diameter measured under a mesopic condition 15 minutes after the sitting position following interscalene brachial plexus block
Post-anesthetic ipsilateral pupil diameter | 30 minutes after interscalene brachial plexus block
  Ipsilateral pupil diameter measured under a mesopic condition 30 minutes after interscalene brachial plexus block
Post-anesthetic contralateral pupil diameter | 30 minutes after interscalene brachial plexus block
  Contralateral pupil diameter measured under a mesopic condition 30 minutes after interscalene brachial plexus block
Pre-anesthetic ipsilateral pupil diameter | 15 minutes after baseline acclimation
  Ipsilateral pupil diameter measured under a mesopic condition 15 minutes after baseline acclimation
Pre-anesthetic contralateral pupil diameter | 15 minutes after baseline acclimation
  Contralateral pupil diameter measured under a mesopic condition 15 minutes after baseline acclimation
Post-sitting parasympathetic nervous activity | 15 minutes after the sitting position following interscalene brachial plexus block
  Natural-log transformed high frequency power of heart rate variability calculated using R wave to R wave intervals obtained for 5 minutes between 10 and 15 minutes after the sitting position following interscalene brachial plexus block
Post-sitting sympathovagal balance | 15 minutes after the sitting position following interscalene brachial plexus block
  Low-to-high frequency power ratio of heart rate variability obtained for 5 minutes between 10 and 15 minutes after the sitting position following interscalene brachial plexus block
Post-sitting overall variability of autonomic nervous system | 15 minutes after the sitting position following interscalene brachial plexus block
  Natural-log transformed total power of heart rate variability obtained for 5 minutes between 10 and 15 minutes after the sitting position following interscalene brachial plexus block
Post-anesthetic sympathetic nervous activity | Between 25 and 30 minutes after interscalene brachial plexus block
  Natural-log transformed low frequency power of heart rate variability between 25 and 30 minutes after interscalene brachial plexus block
Post-anesthetic parasympathetic nervous activity | Between 25 and 30 minutes after interscalene brachial plexus block
  Natural-log transformed high frequency power of heart rate variability between 25 and 30 minutes after interscalene brachial plexus block
Post-anesthetic sympathovagal balance | Between 25 and 30 minutes after interscalene brachial plexus block
  Low-to-high frequency power ratio of heart rate variability between 25 and 30 minutes after interscalene brachial plexus block
Post-anesthetic overall variability of autonomic nervous system | Between 25 and 30 minutes after interscalene brachial plexus block
  Natural-log transformed total power of heart rate variability between 25 and 30 minutes after interscalene brachial plexus block
Pre-anesthetic sympathetic nervous activity | 15 minutes after baseline acclimiation
  Natural-log transformed low frequency power of heart rate variability 15 minutes after baseline acclimation
Pre-anesthetic parasympathetic nervous activity | 15 minutes after baseline acclimiation
  Natural-log transformed high frequency power of heart rate variability 15 minutes after baseline acclimation
Pre-anesthetic sympathovagal balance | 15 minutes after baseline acclimiation
  Low-to-high frequency power ratio of heart rate variability 15 minutes after baseline acclimation
Pre-anesthetic overall variability of autonomic nervous system | 15 minutes after baseline acclimation
  Natural-log transformed total power of heart rate variability 15 minutes after baseline acclimation
Sensory blockade | 30 minutes after interscalene brachial plexus block
  C5 to T1 dermatomal blockade of the shoulder graded from 0 to 2 (0 = no cold sensation, 1 = reduced cold sensation, and 2 = normal cold sensation) by applying ice to the shoulder
Motor blockade | 30 minutes after interscalene brachial plexus block
  Motor blockade of the radial, ulnar, median, musculocutaneous, and axillary nerves graded from 0 to 2 (0 = no block 1 = partial block, and 2 = complete block)

CONTACTS AND LOCATIONS:
Overall Officials: Jong Hae Kim, MD, Principal Investigator — Daegu Catholic University Medical Center
Locations (1):
- Daegu Catholic University Medical Center, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No